CLINICAL TRIAL: NCT03147573
Title: Validity of 1-hour Blood Pressure Monitoring Against the Usual Methods for Diagnosis of Hypertension
Brief Title: Validity of 1BPM for Diagnosis of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci d'Atenció Primària de Salut de l'Eixample (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Dr. Antoni Siso Almirall, Head of Research, Consorci d'Atenció Primària de Salut de l'Eixample
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI16/00660
Record Dates: First submitted 2017-05-02; First posted 2017-05-10 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure monitoring
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood pressure monitoring (Experimental)
  Interventions: Diagnostic Test: 1-hour blood pressure monitoring (1BPM); Diagnostic Test: 24-hour ambulatory blood pressure monitoring (ABPM); Diagnostic Test: Office blood pressure measurement (OBPM); Diagnostic Test: Home blood pressure monitoring (HBPM)

INTERVENTIONS:
Diagnostic Test: 1-hour blood pressure monitoring (1BPM) — This method consists of performing blood pressure measurements programmed at 5-min intervals over 1 hour. Two extra recordings taken at the start and end of this period are discarded. Blood pressure is measured in a quiet room at the same health centre.
Diagnostic Test: 24-hour ambulatory blood pressure monitoring (ABPM) — The device is programmed to record the participant's BP every 20 min and 30 min during the day and night, respectively. Participants are advised to carry on with their normal daily activities, avoiding any intense physical exertion, and to remain at rest when their BP is being measured.
Diagnostic Test: Office blood pressure measurement (OBPM) — Two readings were made one minute apart with a validated automatic sphygmomanometer in a sitting position after five minutes of rest. The average of two readings is calculated. The procedure is repeated during 3 office visits at least a week apart.
Diagnostic Test: Home blood pressure monitoring (HBPM) — For each blood pressure recording, at least two consecutive measurements should be taken, at least one minute apart. Blood pressure should be recorded twice daily, ideally in the morning and evening. Blood pressure recording should continue for at least four consecutive days, ideally seven. The average of the above readings should be calculated, ignoring the first day.

SUMMARY:
Blood pressure measurement methods and conditions are determinants of hypertension diagnosis. The classical methods such as office blood pressure measurement (OBPM) and home blood pressure monitoring (HBPM) have significant limitations. A recent British guideline recommends systematic 24-hour ambulatory blood pressure monitoring (ABPM). However, these devices are not available at all health centers and they can only be used by one patient per day. The aim this study is to validate a new method, 1-hour blood pressure monitoring (1BPM), to diagnose the hypertension.

Participants with suspected hypertension will be recruited from a population of patients seen at three primary health centers in an urban area. According to the sample size estimation, a minimum sample size of 214 participants would be needed for the study. Four diagnostic tests will be performed: OBPM at three visits, HBPM, AMPM and 1BPM. The test order for the 24-hour monitoring, and 1-hour monitoring, will be set randomly. Daytime records of ABPM will be compared to all other monitoring methods using the correlation coefficients and Bland Altman plots. The Kappa index will be used to calculate degree of agreement. The sensitivity and specificity of the methods will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* To visit routinely in the health centres where the study is carried out

Exclusion Criteria:

* Severe physical or cognitive limitations
* Atrial fibrillation or other heart rhythm disorders that could interfere with readings
* Arm Circumference > 42cm
* Arm with arteriovenous fistula
* Mental disorders
* Intolerance to the method of measurement
* Hospitalization during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
1-hour blood pressure monitoring | Assessed at 1 study visit (1 hour)
  Blood pressure measurements obtained by 1-hour blood pressure monitoring
24-hour ambulatory blood pressure monitoring | Assessed at 1 day
  Blood pressure measurements obtained by 24-hour ambulatory blood pressure monitoring
Office blood pressure measurement | Assessed at 3 study visits in two weeks
  Blood pressure measurements obtained by office blood pressure measurement
Home blood pressure monitoring | Assessed twice daily, ideally in the morning and evening, during at least four consecutive days, ideally seven
  Blood pressure measurements obtained by home blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Sisó Almirall, MD PhD, Principal Investigator — Consorci d'Atenció Primària de Salut Barcelona Esquerra (CAPSBE); Luis González de Paz, PhD, Study Chair — Consorci d'Atenció Primària de Salut Barcelona Esquerra (CAPSBE); Belchin Kostov, PhD, Study Chair — Transversal Group for Research in Primary Care, IDIBAPS; Cristina Sierra Benito, MD PhD, Study Chair — Hospital Clinic of Barcelona; Josep Miquel Sotoca, PhD, Study Chair — Hospital Clinic of Barcelona; Mª Carme Alvira, RN, Study Chair — Consorci d'Atenció Primària de Salut Barcelona Esquerra (CAPSBE); Cristina Colungo, RN, Study Chair — Consorci d'Atenció Primària de Salut Barcelona Esquerra (CAPSBE); Berta de Andrés, RN, Study Chair — Consorci d'Atenció Primària de Salut Barcelona Esquerra (CAPSBE); Noemí García, RN, Study Chair — Consorci d'Atenció Primària de Salut Barcelona Esquerra (CAPSBE); Silvia Roura, RN, Study Chair — Consorci d'Atenció Primària de Salut Barcelona Esquerra (CAPSBE)
Locations (3):
- Spain (3):
  - Primary Care Center Les Corts, Barcelona, Catalonia
  - Primary Care Center Casanova, Barcelona, Catalonia
  - Primary Care Center Comte Borrell, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banegas JR, Graciani A, de la Cruz-Troca JJ, Leon-Munoz LM, Guallar-Castillon P, Coca A, Ruilope LM, Rodriguez-Artalejo F. Achievement of cardiometabolic goals in aware hypertensive patients in Spain: a nationwide population-based study. Hypertension. 2012 Oct;60(4):898-905. doi: 10.1161/HYPERTENSIONAHA.112.193078. Epub 2012 Sep 4. PMID 22949530
- [Background] Yang Q, Cogswell ME, Flanders WD, Hong Y, Zhang Z, Loustalot F, Gillespie C, Merritt R, Hu FB. Trends in cardiovascular health metrics and associations with all-cause and CVD mortality among US adults. JAMA. 2012 Mar 28;307(12):1273-83. doi: 10.1001/jama.2012.339. Epub 2012 Mar 16. PMID 22427615
- [Background] Sicras-Mainar A, Navarro-Artieda R. [Cost of arterial hypertension according to levels of morbidity in primary care setting]. Med Clin (Barc). 2009 Sep 5;133(8):290-5. doi: 10.1016/j.medcli.2009.05.017. Epub 2009 Jul 10. Spanish. PMID 19596366
- [Background] ESH/ESC Task Force for the Management of Arterial Hypertension. 2013 Practice guidelines for the management of arterial hypertension of the European Society of Hypertension (ESH) and the European Society of Cardiology (ESC): ESH/ESC Task Force for the Management of Arterial Hypertension. J Hypertens. 2013 Oct;31(10):1925-38. doi: 10.1097/HJH.0b013e328364ca4c. No abstract available. PMID 24107724
- [Background] Piper MA, Evans CV, Burda BU, Margolis KL, O'Connor E, Whitlock EP. Diagnostic and predictive accuracy of blood pressure screening methods with consideration of rescreening intervals: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2015 Feb 3;162(3):192-204. doi: 10.7326/M14-1539. PMID 25531400
- [Background] Krause T, Lovibond K, Caulfield M, McCormack T, Williams B; Guideline Development Group. Management of hypertension: summary of NICE guidance. BMJ. 2011 Aug 25;343:d4891. doi: 10.1136/bmj.d4891. No abstract available. PMID 21868454
- [Background] Siu AL; U.S. Preventive Services Task Force. Screening for high blood pressure in adults: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2015 Nov 17;163(10):778-86. doi: 10.7326/M15-2223. Epub 2015 Oct 13. PMID 26458123
- [Background] Turner JR, Viera AJ, Shimbo D. Ambulatory blood pressure monitoring in clinical practice: a review. Am J Med. 2015 Jan;128(1):14-20. doi: 10.1016/j.amjmed.2014.07.021. Epub 2014 Aug 12. PMID 25107387
- [Background] Chrubasik S, Droste C, Glimm E, Black A. Comparison of different methods of blood pressure measurements. Blood Press Monit. 2007 Jun;12(3):157-66. doi: 10.1097/MBP.0b013e3280ad4073. PMID 17496465
- [Background] Mutlu S, Sari O, Arslan E, Aydogan U, Doganer YC, Koc B. Comparison of ambulatory blood pressure measurement with home, office and pharmacy measurements: is arterial blood pressure measured at pharmacy reliable? J Eval Clin Pract. 2016 Feb;22(1):40-45. doi: 10.1111/jep.12424. Epub 2015 Aug 24. PMID 26303331
- [Background] Gaborieau V, Delarche N, Gosse P. Ambulatory blood pressure monitoring versus self-measurement of blood pressure at home: correlation with target organ damage. J Hypertens. 2008 Oct;26(10):1919-27. doi: 10.1097/HJH.0b013e32830c4368. PMID 18806615
- [Background] Viera AJ, Hinderliter AL, Kshirsagar AV, Fine J, Dominik R. Reproducibility of masked hypertension in adults with untreated borderline office blood pressure: comparison of ambulatory and home monitoring. Am J Hypertens. 2010 Nov;23(11):1190-7. doi: 10.1038/ajh.2010.158. Epub 2010 Jul 29. PMID 20671718
- [Background] Banegas JR, Segura J, Sobrino J, Rodriguez-Artalejo F, de la Sierra A, de la Cruz JJ, Gorostidi M, Sarria A, Ruilope LM; Spanish Society of Hypertension Ambulatory Blood Pressure Monitoring Registry Investigators. Effectiveness of blood pressure control outside the medical setting. Hypertension. 2007 Jan;49(1):62-8. doi: 10.1161/01.HYP.0000250557.63490.55. Epub 2006 Oct 30. PMID 17075026
- [Background] Little P, Barnett J, Barnsley L, Marjoram J, Fitzgerald-Barron A, Mant D. Comparison of agreement between different measures of blood pressure in primary care and daytime ambulatory blood pressure. BMJ. 2002 Aug 3;325(7358):254. doi: 10.1136/bmj.325.7358.254. PMID 12153923
- [Background] Gorostidi M, Banegas JR, de la Sierra A, Vinyoles E, Segura J, Ruilope LM. Ambulatory blood pressure monitoring in daily clinical practice - the Spanish ABPM Registry experience. Eur J Clin Invest. 2016 Jan;46(1):92-8. doi: 10.1111/eci.12565. Epub 2015 Dec 23. PMID 26541761
- [Background] Huckvale C, Car J, Akiyama M, Jaafar S, Khoja T, Bin Khalid A, Sheikh A, Majeed A. Information technology for patient safety. Qual Saf Health Care. 2010 Aug;19 Suppl 2:i25-33. doi: 10.1136/qshc.2009.038497. PMID 20693213
- [Background] van der Wel MC, Buunk IE, van Weel C, Thien TA, Bakx JC. A novel approach to office blood pressure measurement: 30-minute office blood pressure vs daytime ambulatory blood pressure. Ann Fam Med. 2011 Mar-Apr;9(2):128-35. doi: 10.1370/afm.1211. PMID 21403139
- [Background] Mas-Heredia M, Moles-Moliner E, Gonzalez-de Paz L, Kostov B, Ortiz-Molina J, Mauri-Vazquez V, Menacho-Pascual I, Cararach-Salami D, Sierra-Benito C, Siso-Almirall A. Validity and applicability of a new recording method for hypertension. Rev Esp Cardiol (Engl Ed). 2014 Sep;67(9):717-23. doi: 10.1016/j.rec.2013.12.017. Epub 2014 Apr 30. PMID 25172067
- [Derived] Siso-Almirall A, Kostov B, Blat E, Garcia N, de Andres B, Roura S, Sierra-Benito C, Alvira-Balada MC, Colungo C, Benavent-Areu J, Gonzalez-de Paz L. Validity and reliability of 1-h automated office blood pressure measurement for the diagnosis of hypertension. J Hypertens. 2022 Mar 1;40(3):453-461. doi: 10.1097/HJH.0000000000003029. PMID 34654792
- [Derived] Gonzalez-de Paz L, Kostov B, Alvira-Balada MDC, Colungo C, Garcia N, Roura S, Blat E, Sierra-Benito C, Sotoca-Momblona JM, Benavent-Areu J, Sanchez E, Siso-Almirall A; Eva Sanchez on behalf of the OMBP Group. Effectiveness of a new one-hour blood pressure monitoring method to diagnose hypertension: a diagnostic accuracy clinical trial protocol. BMJ Open. 2019 May 27;9(5):e029268. doi: 10.1136/bmjopen-2019-029268. PMID 31133597